CLINICAL TRIAL: NCT05652062
Title: An Exploratory Study to Evaluate the Prizvalve® System in Patients With Failing Bioprosthetic Valve
Brief Title: Prizvalve® Transcatheter Valve-in-Valve Implantation Exploratory Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai NewMed Medical Co., Ltd. (Industry)
Collaborators: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Prizvalve-VIV-2022
Record Dates: First submitted 2022-12-08; First posted 2022-12-15 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Failing Bioprosthetic Valve

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Device: Prizvalve® system

INTERVENTIONS:
Device: Prizvalve® system — Transcatheter valve-in-valve replacement

SUMMARY:
The primary purpose of this clinical trial is to evaluate the efficacy and safety of the transcatheter aortic valve system in the treatment of patients with failing bioprosthetic valve

DETAILED DESCRIPTION:
The Prizvalve® study is a single-center, single-arm, prospective, exploratory clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Failing bioprosthetic valve (≥moderate stenosis and/or ≥moderate regurgitation);
2. Age≥18 years old who are not in pregnancy or lactation;
3. NYHA Function Class≥ II;
4. Patient who is anatomically suitable for the implantation of the Prizvalve® ;
5. According to heart team , patient is intermediate or above surgical risk or not suitable for redo open heart surgery of valve replacement due to other severe comorbidities ;
6. Heart team agrees valve implantation will likely benefit the patient;
7. Patient understands the purpose of the trial and volunteers to participate in, sign the informed consent form and is willing to accept relevant examinations and clinical follow-ups.

Exclusion Criteria:

1. Patients with other valvular diseases that require simultaneous intervention;
2. Patients with other heart diseases that require simultaneous intervention;
3. Estimated life expectancy < 12 months;
4. Failing valve has moderate and above paravalvular regurgitation;
5. Failing valve in unstable ore not structurally intact;
6. Increased risk of coronary artery obstruction by prosthetic leaflets of the failing valve;
7. Anatomical characteristics that would preclude transcatheter valve implantation;
8. Anatomical characteristics that would increase the risk of left ventricular outflow tract (LVOT) obstruction;
9. Patient with acute myocardial infarction within 30 days;
10. Any therapeutic cardiac operation (excluding previous PCI and pacemaker implantation) is performed within 30 days of the index procedure;
11. Patient with hypertrophic cardiomyopathy with obstruction;
12. Echocardiographic evidence of intracardiac mass, thrombus or vegetation;
13. Patients with active infective endocarditis or other active infections;
14. Patients with severe right ventricular dysfunction, or severe left ventricular dysfunction, left ventricular ejection fraction (LVEF) < 20%;
15. Patients who cannot tolerate anticoagulant or antiplatelet therapy;
16. Patients with severe untreated coronary artery stenosis requiring revascularization;
17. Patients with cerebrovascular accident within 3 months, excluding transient ischemic attack;
18. Patients who refuse surgical treatment in emergency situations under any circumstances;
19. Patients who have severely disabled Alzheimer's disease and inability to take care of themselves;
20. Patients who have participated in clinical trials of other drugs or medical devices before enrollment and have not yet reached the primary outcome of research;
21. The investigator judged that patient with poor compliance and could not complete the study as required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2022-06-02 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06-02 (Estimated)

PRIMARY OUTCOMES:
Composite of all-cause mortality and valve-related reintervention | 1 year

SECONDARY OUTCOMES:
Technical success | 30 days
  1. Freedom from death;
  2. Successful vascular delivery and retrieval of transcatheter valve delivery system;
  3. Correct position of transcatheter valve;
  4. No need for any emergency surgery or re-intervention (including device-related and surgical approach-related);
  5. Adequate performance of prosthesis (No moderate or greater stenosis or regurgitation).
Procedural Success | 30 days
  1. Device success;
  2. No severe complications of the following: death; stroke; life threatening bleeding; major vascular complications; secondary severe cardiac organic disease (eg: aortic dissection, apical aneurysm formation, left ventricular outflow tract obstruction, etc.); stage 2 or 3 AKI; MI or coronary ischemia requiring PCI or CABG; severe hypotension; heart failure or respiratory failure requiring high-dose vasoactive drugs/or cardiac mechanical assist devices; any valve-related dysfunction including migration, thrombosis, or other complication requiring surgery or repeat intervention.
Device success | 30 days
  1. Freedom from stroke;
  2. Prosthetic heart valve function is normal (including no displacement, calcification, thrombosis, hemolysis, or endocarditis);
  3. No need for any emergency surgery or secondary intervention (including device-related and surgical approach-related);
  4. No prosthetic valve stenosis；
  5. Prosthetic valve regurgitation <2+ (including central leakage and paravalvular leakage), and no related hemolysis;
  6. LVOT pressure gradient increased <20mmHg.
All-cause mortality | 30 days
  All-cause mortality included cardiac，non-cardiac death and other ominous death.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China